CLINICAL TRIAL: NCT04058678
Title: Effects of Telomerase Reactivation With Danazol in Ovarian Function.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, Juan A Garcia-Velasco, PhD in Medicine and gynecology, University professor, IVI Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1707-FIVI-084-MV
Record Dates: First submitted 2019-08-12; First posted 2019-08-15 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Ovarian Reserve
Keywords: Ovarian reserve.; Telomeric factor; Blood; Granulosa cells
MeSH Terms: interventions — Danazol; Methods

STUDY DESIGN:
Intervention Model Description: A control group composed of women with normal ovarian reserve to compare telomeric and fertility parameters with the group with compromised ovarian reserve.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the first visist to the doctor, women will be selected according to the selection criteria. Those who seem to have a low ovarian reserve by ultrasound will be informed of the trial, and if they decide to participate, blood will be taken to analyze AMH values. On the second visit, women with low ovarian reserve will be randomized 1:1 for either inactive substance or Danazo, accordint to a computer-generated randomization list prepared by associated statistic. This way, the assigned group will be blind until the momento of executing the randomization procedure. Moment in which, the assigned group will be revealed.
  Those with normal ovarian reserve will not be randomized and will just be included as controls.
  To maintain the blinding of the trial, Danazol and placebo will be provided in boxs with blisters (PVC opaque and aluminium sealed).
  Only the trial medication delegate(s) at the site will dispense the IMP and will know the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (Sham Comparator): A control group composed of women with normal ovarian reserve (30 to 45 yerras old) is needed to compare telomeric and fertility parameters with the group of women with compromised ovarian reserve. Note that the term "normal ovarian reserve" referred to older women indicates women that still have follicles in their ovaries -and thus, normal AMH values-, even though the number may be lower tan at a younger age or the quality of oocytes may be lower tan in younger women. In other words, women in the control group irrespective of their age, will have a greater number of follicles compared to women belonging to the group with compromised ovarian reserve.
  Interventions: Other: Without intervention
- EXPERIMENTAL (Experimental): A group of women with diminished ovarian reserve that will take an inactive substance has been included to avoik biases and to set the fertility base line for women with compromised ovarian reserve.
  Interventions: Drug: Danazol/Placebo

INTERVENTIONS:
Drug: Danazol/Placebo — This group will be randomized 1:1 for either inactive substance or Danazol, according to a computer-generated randomization list prepared. Women will be treated with Danazol/Placebo oral way for 3 months.
  Arms: EXPERIMENTAL
Other: Without intervention — Women with normal ovarian reserve will not be treated in anyway, thus, randomization will not be necessary.
  Arms: CONTROL

SUMMARY:
This project explores the implication of the telomere pathway in ovarian premature and regular aging. Telomere length and maintenance underlie several biological processes such cancer, aging, human diseases and the biology of stem cells. The reactivation of telomerase should lead to a rejuvenation of the ovarian tissue and the improvement of fertility.

The correlation of telomeric factors in blood and granulosa cells will be studied with the aim of finding telomeric biomarkers of ovarian aging.

DETAILED DESCRIPTION:
This is a pilot study, randomized, controled, blind, parallelo arm clinical trial with inactive substance and medicine.

A pilot study will be developed with a total of 45 individuals from 30 to 45 years old, who represent the most frequent population of women seeking for ART.

A control group composed of women with normal ovarian reserve (30 to 45 years old) is needed to compare telomeric and fertility parameters with the group of women with compromised ovarian reserve. Women in the control group irrespective of their age, will have a greater number of follicles compared to women belonging to the group with compromised ovarian reserve.

A group of women with diminished ovarian reserve that will take an inactive substance has been incluided to avoid biases and to set the fertility base line for women with compromised ovarian reserve. The use of an inactive substance or placebo will help obtain better quality results. For instance, if Danazol happened to improve the fertility outcome, then, there could be a possibility that the IVF improvement might be due to other components of the pill. Using placebo, this possibility would be eliminated, since the placebo will contain all components of the pill, except Danazol.

The development of a pilot study will help us understand the statisticl behavior or the telomeric factors as well as to determine the appropriate number of individuals that shoyuld be recruited in a clinical trial to have results with statistical significance. In addition, a pilot study will help us learn errors or undesired events that may happen during the clinical trial. For instance, if patients cannot follow the indications of their doctors and why, or what proportion of patients will drop the study and the reasons for it. Furthermore, it will also help us understand if there exist a tendency, an indication or even a clear beneficial effect for patients without harming them.

The number of participants selected for the study is considered adequate for each group, since each group will be measured in an independent manner.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of the study. This include the decisión to use contraception methods different to sexual hormones, such as the use of condoms, during the treatment with Danazol.
* In good general health as evidenced by medical history or diagnosed with body mass index between 18 and 30 kg/m2.
* Women with normal (AMH valued must be equal or higher tan 2ng/ml) or compromised ovarian reserve (defined as AMH < 2 ng/ml)
* Not having had any steroid hormones for one month.

Exclusion Criteria:

* Pregnancy o lactation.
* Taking other sexual hormones.
* Women with diseases in heart, liver or kidney or tumors which depend on male sexual hormones or hormone-dependent tumour.
* Women taking anticonvulsants, medicaments for diabetes, anticoagulants and anti-hypertension: ciclosporin and tacrolimus and other steroids and statins.
* Women suffering irregular genital bleeding or with thrombus or thromboembolicdiseases.
* Known allergic reactions to components of the study product (cornstarch and lactose).
* Having received ovulation induction drugs within one month before the inclusión in the study.
* Anything that would place the individual at increased risk or preclude the individual´s full compliance with or completion of the study.
* Simultaneous participation in another clinical trial or previous participation in this study.
* Participation in another clinical study 2 months before inclusión in the present study that could affect its objectives.

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Most frequent population of women seeking for ART
Enrollment: 19 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Telomere length in granulosa cells | The evaluation of the main assessment criterion will be done both after eighth visit (36 hours post induction) for women with low ovarian reserve and fifth visit for woman with normal ovarian reserve
  Measured in arbitrary units of fluorescence (a.u.) from 0 to 255 gray intensity (8bit) or Kb (continuous variable). Below 3 kb are considered critically short telomeres in humans.

SECONDARY OUTCOMES:
Accumulation of short telomeres | Through study completion, an average of 1 year
  Measured in arbitrary units of fluorescence (a.u.) from 0 to 255 gray intensity (8bit) or Kb (continuous variable). Below 3 kb are considered critically short telomeres in humans.
Telomerase activity | Through study completion, an average of 1 year
  Product of PCR amplification, run in acrylamide gels and quantified as band intensity (continuous variable)
DNA damage measurement | Through study completion, an average of 1 year
  If damage is positive, then different foci should be apparent in the nucleus of the cell. The number of foci present in the nuclei of at least 100 cells will be counted. If there is DNA damage at telomeres, then yH2AX or 53BPI foci will colocalize with telomeres (labelled with anti TRF1 antibody). Spots will be counted (continuous variable).
Other telomeric factors. | Through study completion, an average of 1 year
  The mRNA expression levels of the telomerase gene and the shelterins, which are involved in telomere lengthening and protection, will be measured by qPCR. (continuous variable).

CONTACTS AND LOCATIONS:
Overall Officials: María Elisa Varela, Principal Investigator — IVIRMA MADRID
Locations (1):
- Ivirma Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armanios MY, Chen JJ, Cogan JD, Alder JK, Ingersoll RG, Markin C, Lawson WE, Xie M, Vulto I, Phillips JA 3rd, Lansdorp PM, Greider CW, Loyd JE. Telomerase mutations in families with idiopathic pulmonary fibrosis. N Engl J Med. 2007 Mar 29;356(13):1317-26. doi: 10.1056/NEJMoa066157. PMID 17392301
- [Background] Blasco MA, Lee HW, Hande MP, Samper E, Lansdorp PM, DePinho RA, Greider CW. Telomere shortening and tumor formation by mouse cells lacking telomerase RNA. Cell. 1997 Oct 3;91(1):25-34. doi: 10.1016/s0092-8674(01)80006-4. PMID 9335332
- [Background] Blasco MA. Telomeres and human disease: ageing, cancer and beyond. Nat Rev Genet. 2005 Aug;6(8):611-22. doi: 10.1038/nrg1656. PMID 16136653
- [Background] Bernardes de Jesus B, Vera E, Schneeberger K, Tejera AM, Ayuso E, Bosch F, Blasco MA. Telomerase gene therapy in adult and old mice delays aging and increases longevity without increasing cancer. EMBO Mol Med. 2012 Aug;4(8):691-704. doi: 10.1002/emmm.201200245. Epub 2012 May 15. PMID 22585399